CLINICAL TRIAL: NCT01559519
Title: Effect of Albumine Infusion in the Prevention of Hepatic Encephalopathy After Transjugular Intrahepatic Portosystemic Shunt
Brief Title: Post Transjugular Intrahepatic Portosystemic Shunt (Tips) Albumine Infusion to Prevent Hepatic Encephalopathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Prof oliviero Riggio, Professor, University of Roma La Sapienza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2012-000931-20
Record Dates: First submitted 2012-03-06; First posted 2012-03-21 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Hepatic Encephalopathy
Keywords: TIPS; albumin; hepatic encephalopathy; hyponatremia; hypovolemia; cirrhosis
MeSH Terms: conditions — Hepatic Encephalopathy; Hyponatremia; Hypovolemia; Fibrosis | interventions — Albumins; Serum Albumin, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- albumin (Active Comparator): cirrhotic patients who underwent tips placement
  Interventions: Drug: Albumin

INTERVENTIONS:
Drug: Albumin — albumin 20% 1 g/Kg body weight for the first two days after TIPS followed by 0,5 g/Kg body weight at day 4 and then 0,5 g/Kg body weight once a week for three weeks.
  Other Names: human albumin

SUMMARY:
The purpose of this study is to evaluate the efficacy of albumin infusion to prevent post tips hepatic encephalopathy'

DETAILED DESCRIPTION:
The outcome is the prevention of post tips hepatic encephalopathy

ELIGIBILITY:
Inclusion Criteria:

* Cirrhotic patients
* TIPS placement
* Absence of Hepatic Encephalopathy at the enrolement
* Age > 18 years
* No pregnancy

Exclusion Criteria:

* Non-cirrhotic portal hypertension
* Previous liver transplantation
* Impossibility to attend the scheduled follow-up including the weekly visit as outpatients during the first month after TIPS (see the description of follow-up below)
* Sings of overt hepatic encephalopathy as well as a history of persistent HE at entry. The latter as a contraindication for TIPS placement

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
one or more episodes of hepatic encephalopathy (> grade 2 according to West Heven criteria)after TIPS placement | one month post tips
  evaluate the efficacy of albumin infusion to prevent the occurrence of hepatic encephalopathy (> grade 2 according to West Heven criteria)one months after tips placement

SECONDARY OUTCOMES:
arterial blood pressure >120/80 mmHg and natremia >130 mg/dl in cirrhotic patients one month after TIPS placement | one month after tips placement
  improving the hypovolemia, evaluated by the arterial blood pressure value, and hyponatremia (<130 mg/dl)after albumine infusion for one month after tips placement

CONTACTS AND LOCATIONS:
Overall Officials: oliviero riggio, professor, Principal Investigator — University of Roma La Sapienza